CLINICAL TRIAL: NCT00615173
Title: Prospective, Randomized, Multicenter, Control Study to Assess the Efficacy and Safety of Tacrolimus in Induction and Maintenance Phase Treatment in Lupus Nephritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Xueqing Yu, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSU-PRGLN-001
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Kidney Diseases; Lupus Nephritis; Tacrolimus; Induction Phase; Maintenance Phase
Keywords: Tacrolimus; lupus nephritis
MeSH Terms: conditions — Kidney Diseases; Lupus Nephritis | interventions — Tacrolimus; Cyclophosphamide; Azathioprine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): tacrolimus(fk506) treatment in induction and maintenance phase
  Interventions: Drug: tacrolimus (FK506)
- 2 (Active Comparator): intravenous cyclophosphamide pulses treatment in induction phase; and Aza in the maintenance phase
  Interventions: Drug: cyclophosphamide or azathioprine

INTERVENTIONS:
Drug: tacrolimus (FK506) — Started: 0.05-0.1mg/kg/d,divided into two daily dose at 12hr; the blood level:5-10ng/ml in induction phase;and 4-6ng/ml in maintenance phase;
  Arms: 1
Drug: cyclophosphamide or azathioprine — Induction phase: CTX 0.75g/m2 monthly Maintenance phase: AZA 2mg/kg/d.
  Arms: 2

SUMMARY:
The purpose of this study is to compare the efficacy and safety of tacrolimus vs intravenous cyclophosphamide pulses treatment for the induction therapy of LN(III,IV,V).

To compare the efficacy and safety of tacrolimus vs Azathioprine for the maintenance therapy of LN(III,IV,V).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects of either sex, 14-65 years of age;
2. Diagnosis of SLE according to the ACR criteria(1997);
3. Kidney biopsy within the 6 months prior to first randomization with a histologic diagnosis (ISN/RPS 2003 classification of LN) class III, IV, V;
4. Class IV LN: proteinuria >1g/24hr or Scr>115umol/L;
5. Class III or V LN: proteinuria >2g/24hr or Scr>115umol/L;
6. Provision of written informed consent by subject or guardian.

Exclusion Criteria:

1. Inability or unwillingness to provide written informed consent ;
2. Known hypersensitivity or contraindication to tacrolimus, cyclophosphamide , azathioprine, corticosteroids;
3. Usage of immunosuppression therapy (MMF, CTX, CysA, MTX ect) for more than 1 week within 1 month prior to first randomization;
4. Pregnancy, nursing or use of a non-reliable method of contraception;
5. Continuous dialysis starting more than 2 weeks before randomization into the induction phase and/or continuous dialysis with an anticipated duration of more than 8 weeks;
6. Previous kidney transplant or planted transplant;
7. Scr > 4mg/dl (353umol/L);
8. Active hepatitis, with liver dysfunction;
9. Diagnosed DM;
10. Participation in another clinic trial and/or receipt of investigational drugs within 4 weeks prior to screening .

Ages: 14 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2006-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Remission rate | 2006-2008

SECONDARY OUTCOMES:
Renal function, proteinuria, relapse. | 2006-2008

CONTACTS AND LOCATIONS:
Overall Officials: Xue Qing Yu, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital, Sun Yat-Sen University; Ping Fu, MD, Principal Investigator — Department of Nephrology, West China Hospital of Sichuan University; Yun Hua Liao, MD, Principal Investigator — Department of Nephrology, 1st Affiliated Hospital of Guangxi Medical University; Jin li Zhang, MD, Principal Investigator — Department of nephrology, People's Hospital of Yunnan Province; Jian Chen, MD, Principal Investigator — Department of Nephrology, Fuzhou Military General Hospital; Tan Qi Lou, MD, Principal Investigator — Department of Nephrology, 3rd Affiliated Hospital of Sun Yet-Sen University; Yao zhong Kong, MD, Principal Investigator — Department of Nephrology, 1st People's Hospital of Foshan; Jun zhou Fu, MD, Principal Investigator — Department of Nephrology,1st People's Hospital of Guangzhou; Wei Shi, MD, Principal Investigator — Department of Nephrology, People's Hospital Guangdong Provincial; Zheng rong Liu, MD, Principal Investigator — Department of Nephrology, Nanfang Hospital of Southern Medical University
Locations (1):
- The 1st Affiliated Hospital, Sun Yet-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Chen W, Tang X, Liu Q, Chen W, Fu P, Liu F, Liao Y, Yang Z, Zhang J, Chen J, Lou T, Fu J, Kong Y, Liu Z, Fan A, Rao S, Li Z, Yu X. Short-term outcomes of induction therapy with tacrolimus versus cyclophosphamide for active lupus nephritis: A multicenter randomized clinical trial. Am J Kidney Dis. 2011 Feb;57(2):235-44. doi: 10.1053/j.ajkd.2010.08.036. Epub 2010 Dec 21. PMID 21177013